CLINICAL TRIAL: NCT01057784
Title: Bariatric Surgery Outcomes: Quality of Life / Reproductive-Age Women
Brief Title: Bariatric Surgery Outcomes
Status: Withdrawn | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Daniel DeUgarte, MD, UCLA
Other Study IDs: 09-11-095
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2010-01

CONDITIONS: Morbid Obesity
Keywords: obesity; bariatric; surgery; sleeve; gastric bypass; vitamin D; quality of life; body composition; bone density; adolescent; child; teenager; fertility; offspring; biomarker; epigenome; gene expression
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The subgroup of 10 reproductive-age women will have coded bloods samples retained for DNA and RNA analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric Surgery Patients: Patients undergoing bariatric surgery.
  Interventions: Procedure: Bariatric surgery.
- Reproductive-Age Women - Bariatric Surgery Patients: This subgroup of patients will include 10 reproductive-age women.
  Interventions: Procedure: Bariatric surgery.

INTERVENTIONS:
Procedure: Bariatric surgery. — Bariatric Surgery

SUMMARY:
The UCLA Metabolic and Bariatric Surgery Program (adult program) and the UCLA Fit for Healthy Weight Program (adolescent program) are committed to the care of morbidly obese patients. This study is observational. The investigators plan to evaluate bariatric surgery outcomes using the BAROS National Database and also to evaluate quality of life pre- and post bariatric surgery. In addition, the investigators plan to enroll a subgroup of 10 reproductive-age women to evaluate: 1) pregnancy and offspring health, 2) long-term nutrition, 3) biomarkers/epigenome, and 4) body-composition/bone-density.

DETAILED DESCRIPTION:
1. National Database: The purpose of the Bariatric Outcomes Longitudinal Database (BOLD) study is to study the mid- and long-term outcomes of bariatric surgeries and to analyze the relationship between these outcomes and 1) patient demographics and comorbidities, 2) clinical and surgical characteristics, and 3) pre-operative, peri-operative, and post-operative care and treatment. The UCLA program will be just one of many institutions that participate in the BOLD study. Participants include other programs and surgeons who have received a Full Approval or Provisional Status designation in the American Society for Bariatric Surgery (ASBS) Bariatric Surgery Center for Excellence program. This study, along with the database itself, is being established, maintained and overseen by East Carolina University in association with the Surgical Review Corporation.
2. Health Survey: The purpose of evaluating physical and mental health is to document changes that occur following surgery. Standardized surveys will include SF-36, (Bariatric Analysis and Reporting Outcome System), BAROS, and Epworth Sleepiness Scale. Our hypothesis is that bariatric surgery will improve quality of life for the majority of patients.
3. Reproductive-Age Women:

While the number of bariatric procedures performed has increased to over 200,000 annually, this number represents only a small fraction of those that qualify. The prevalence of extreme obesity is higher in women than in men (7% vs. 3%), and women are disproportionately more likely to undergo bariatric surgery. Nearly 80% of patients undergoing bariatric surgery are female and 35% are less than 40 years of age.

Given the current demographics of metabolic/bariatric surgery and the epidemic of childhood obesity, it is important to evaluate the long-term impact of bariatric surgery on nutrition, pregnancy, offspring health, and bone density. Despite previous concerns, metabolic/bariatric surgery has been demonstrated to improve maternal outcomes and likely improves neonatal outcomes. Interestingly, weight-loss surgery has been demonstrated to reduce the incidence of obesity in offspring by 50%. It is unclear whether improvements in offspring health are related to changes in the uterine environment, the post-natal environment, or the epigenome.

While obesity has been associated with Vitamin D deficiency and hyperparathyroidism, it is not usually associated with the development of osteoporosis. Bariatric surgery can impair calcium absorption and exacerbate vitamin deficiencies. However, the impact of surgery on bone mineral content and density is unclear. This has particular ramifications for young female patients and the risk of osteoporosis long-term.

The purpose is this portion of the study is to evaluate the impact of metabolic/bariatric surgery on reproductive-age women (age 13 to 30) with respect to weight, nutritional status, body composition, biomarker/epigenome profile, markers of atherosclerosis, and bone mineral content/density.

1. Obstetrical/Offspring Health and Fertility: The purpose of this assessment is to evaluate the impact of surgery on obstetrical complications, offspring health, and fertility. A simple questionnaire will be administered to women of reproductive age.
2. Biomarkers /Epigenetic Markers: The purpose of collecting specimens (e.g. blood) and analyzing changes in hormones, biologic markers, and epigenetic markers is to help elucidate potential mechanism involved in weight loss.
3. Imaging: In collaboration with Children's Hospital - Los Angeles, we will coordinate imaging to evaluate body composition, bone density/content, and subclinical markers of atherosclerosis. Imaging studies will include DEXA (dual x-ray absorptiometry) for patients under 300 lbs, low-dose CT-scan for patients under 350 lbs, and ultrasound of the vessels of the neck.

ELIGIBILITY:
1. Bariatric Surgery Patient Cohort:

   Inclusion Criteria:
   * Patients undergoing bariatric surgery.

   Exclusion Criteria:
   * None
2. Reproductive-Age Women Patient Cohort:

Inclusion Criteria:

* Patients undergoing bariatric surgery.
* Age 13-30 females.
* Weight less than 350lbs (to accommodate imaging).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life. | up to 5-year.
Biomarkers, RNA Expression Profile, Epigenetic Markers | up to 5-year
Bone density/content and body composition. | up to 5-year.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DeUgarte, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital - Los Angeles, Los Angeles, California
  - UCLA, Los Angeles, California

REFERENCES:
- See also: UCLA Fit for Healthy Weight Program — http://fitprogram.ucla.edu
- See also: UCLA Metabolic and Bariatric Surgery Program — http://bariatrics.ucla.edu/